CLINICAL TRIAL: NCT00379717
Title: Concurrent Helical Tomotherapy With Chemotherapy in Unresectable Stage III Non-Small Cell Lung Cancer (NSCLC): a Phase I/II Trial of Radiation Dose Escalation and Fixed Dose Chemotherapy.
Brief Title: Concurrent Helical Tomotherapy With Chemotherapy in Unresectable Stage III Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ-VUB (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Bral Samuel, UZ Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VUB06-001; TomoCT
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2006-09

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: helical tomotherapy; dose escalation; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Drug: Cisplatinum
Drug: Docetaxel
Device: Tomotherapy

SUMMARY:
This non-randomized Phase I/II study is designed to determine the maximum tolerated dose (MTD) of thoracic radiotherapy and concurrent chemotherapy with cisplatin and docetaxel in patients with LA-NSCLC. All patients will receive weekly administrations of docetaxel 20 mg/m² and cisplatin 20 mg/m2 concurrently with radiotherapy. Radiotherapy will be delivered using helical tomotherapy in 30 daily fractions over six weeks. Patients should have recovered fully from induction concurrent chemoradiotherapy before they continue with the consolidation chemotherapy phase. Patients will be entered in cohorts of at least 5 subjects.

The first cohort of patients will receive 30 fractions of 2Gy in six weeks up to a total dose of 60Gy. The concurrent chemotherapy starts at day 1 of the radiotherapy and will be administered 2-4 hours before the radiotherapy.

The radiotherapy fraction size will be escalated to 2.36Gy in three steps.

DETAILED DESCRIPTION:
Dose escalation steps are:

30*2.00Gy = 60.0Gy (BED= 70.8Gy10 NID2= 60.0Gy) 30*2.12Gy = 63.6Gy (BED= 75.9Gy10 NID2= 64.2Gy) 30*2.24Gy = 67.2Gy (BED= 81.5Gy10 NID2= 68.5Gy) 30*2.36Gy = 70.8Gy (BED= 86.3Gy10 NID2= 72.9Gy) If MTD is not reached, protocol modification allowing further escalation can be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent is required.
2. Histologically or cytologically confirmed NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma or a combination of these)
3. Patients must have a stage III unresectable LA-NSCLC:
4. Males or females aged between 18 and 75 years.
5. Life expectancy of at least 12 weeks.
6. ECOG performance status 0,1 or2.
7. Weight loss ≤ 10% within the last 3 months.
8. Laboratory requirements at entry:

   • Blood cell counts: i. Absolute neutrophils ≥ 2.0 x 109/L ii. Platelets ≥ 100 x 109/L iii. Haemoglobin ≥ 11 g/dl

   • Renal function: i. Serum creatinine < 1 x the upper limit of normal (UNL). ii. In case of borderline value of serum creatinine, the 24h creatinine clearance should be > 60 ml/min.

   • Hepatic function: i. Serum bilirubin < 1 x UNL ii. ASAT and ALAT < 2.5 x UNL iii. alkaline phosphatase < 5 x UNL iv. Patient with ASAT and/or ALAT > 1.5 x UNL associated with alkaline phosphatase> 2.5 x UNL is not eligible for the study.
9. Lung function tests at entry:

   * FEV1: ≥ 50 % x Normal value
   * DLCO: ≥ 50 % x Normal value
10. Adequate cardiac function.
11. Patient with either measurable and/or non-measurable lesion (according to RECIST criteria, A1).

Exclusion Criteria:

1. Diagnosis of small cell lung cancer.
2. Stage IIIB NSCLC, based on the presence of malignant pleural or pericardial effusion.
3. Pregnant or lactating women.
4. Patients (male or female) with reproductive potential not implementing adequate contraceptive measures.
5. Prior systemic chemotherapy, immunotherapy, or biological therapy including neoadjuvant or adjuvant treatment for NSCLC.
6. Prior surgery for NSCLC, if less than 5 years from study.
7. Prior radiotherapy for NSCLC.
8. History of prior malignancy, except for cured non-melanoma skin cancer, curatively treated in-situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least five years.
9. Symptomatic peripheral neuropathy Grade ≥ 2 except if due to trauma.
10. Other serious concomitant illness or medical conditions:
11. Congestive heart failure or angina pectoris except if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or arrhythmias.
12. History of significant neurological or psychiatric disorders including dementia or seizures.
13. Active infection requiring IV antibiotics.
14. Active ulcer, unstable diabetes mellitus or other contra-indication to corticosteroid therapy.
15. Superior vena cava syndrome contra-indicating hydration.
16. Pre-existing pericardial effusion.
17. Pre-existing symptomatic pleural effusion.
18. Significant gastrointestinal abnormalities, including requirement for intravenous nutrition, active peptic ulcer disease, prior surgical procedures affecting absorption.
19. Distant metastasis.
20. Concurrent treatment with any other experimental anti-cancer drugs.
21. Concomitant or within 4-week period administration of any other experimental drug under investigation.
22. Significant ophthalmologic abnormalities.
23. Moderate to severe dermatitis.
24. Hypersensitivity to docetaxel, cisplatin, or any of its excipients.
25. Concomitant use of phenytoin, carbamazepin, barbiturates, or rifampicin.
26. Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
27. Patient unlikely to comply with protocol, i.e., uncooperative attitude, inability to return for follow-up visits, and not likely to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-11; Study Completion 2008-04

PRIMARY OUTCOMES:
To evaluate the feasibility and toxicity of radiation dose escalation using helical tomotherapy concurrently with chemotherapy (docetaxel-cisplatin combination) in stage III locally advanced non small cell lung cancer (LA-NSCLC).

SECONDARY OUTCOMES:
To estimate efficacy parameters in terms of overall response rate, progression free survival and overall survival. To monitor quality of life (QOL) before, during and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Bral, MD, Principal Investigator — AZ-VUB
Locations (1):
- UZ Brussel, Jette, Belgium